CLINICAL TRIAL: NCT00185887
Title: Nitroglycerin Versus Terbutaline for Intrapartum Fetal Resuscitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Yasser Yehia El-Sayed, Stanford University School of Medicine
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 79504
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-03

CONDITIONS: Fetal Distress
MeSH Terms: conditions — Fetal Distress | interventions — Terbutaline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Terbutaline (Active Comparator)
  Interventions: Drug: Terbutaline
- Nitroglycerine (Active Comparator)
  Interventions: Drug: Terbutaline

INTERVENTIONS:
Drug: Terbutaline — Terbutaline 250 micrograms intravenously for intrapartum fetal resuscitation. Nitroglycerine 400 micrograms intravenously for intrapartum fetal resuscitation.

SUMMARY:
To compare nitroglycerin and terbutaline for intrapartum fetal heart rate resuscitation

ELIGIBILITY:
Inclusion Criteria::

* nonreassuring fetal heart rate tracing Exclusion Criteria:- maternal cardiac disease, placental abruption, intrauterine growth restriction, prior cesarean section

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2003-10; Primary Completion 2006-07 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
resolution of abnormal fetal heart tracing | Administration of study medication to resolution of abnormal fetal heart tracing or operative delivery.

SECONDARY OUTCOMES:
cesarean section rate | Data analysis
operative vaginal delivery rate | Data analysis
neonatal outcomes | time of delivery to time of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Yehia El-Sayed, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States